CLINICAL TRIAL: NCT04413916
Title: ASSOCIATION OF miRNA WITH ALLOGRAFT FUNCTION AND EXPRESSION PROFILES PREDICTIVE OF DISEASES OCCURING AFTER KIDNEY TRANSPLANTATION
Brief Title: MiRNA in Kidney Transplantation: Association With Kidney Graft Function and Disease Process
Status: Completed | Type: Observational
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Veceric-Haler Zeljka, assist. prof., University Medical Centre Ljubljana
Other Study IDs: P20190104
Record Dates: First submitted 2020-05-25; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-05

CONDITIONS: Kidney Transplant Failure and Rejection
Keywords: miRNA; kidney transplant function; kidney transplant rejection; disease recurrence; cystatin; micro RNA
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Serums from kidney transplant recipients
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: miRNA expression — Analysis of expression of selected miRNAs (miR-29c, miR-126, miR-146a, miR-150, miR-155, miR-223) by qPCR.

SUMMARY:
MicroRNAs (miRNAs) belong to a class of small non-coding RNAs that modulate physiological and pathological processes by post-transcriptional regulation of gene expression mainly via translational inhibition of target messenger RNAs. Recently, many miRNAs were found to be involved in pathological processes that occur following kidney transplantation, like allograft rejection, de novo disease or disease recurrence after kidney transplantation. As most of the miRNAs involved in kidney diseases are extracted by urine, the diagnostic accuracy of such molecules as biomarkers is questionable.

The aim of this study is to analyze expression of selected miRNAs (miR-29c, miR-126, miR-146a, miR-150, miR-155, miR-223) and evaluate whether their regulation is associated with kidney graft function and disease processes after kidney transplantation (KTx).

DETAILED DESCRIPTION:
MicroRNAs (miRNA) are short, endogenous non-coding RNAs involved in the modulation of gene expression mainly by inhibition of messenger RNAs translation. Recent studies have indicated association of miRNAs with pathological processes following kidney transplantation.

The aim of the study is to determine whether selected miRNAs are related to specific disease process or only reflect kidney graft function.

The study enrolled 100 Caucasian KTRs, who presented with stable renal function (as indicated by stable serum creatinine (Cr) for 3 months and whose kidney graft function was thereafter estimated with various methods, including: cystatin C concentration, three different CKD EPI equations and measured with chromium-51 ethylenediamine tetraacetic acid clearance.

Expression of 6 selected miRNAs (miR-29c, miR-126, miR-146a, miR-150, miR-155, and miR-223) was determined by qPCR using miRNA-103a, miR-191, and miR-423 as reference genes.

ELIGIBILITY:
Inclusion criteria:

* time of kidney transplantation at least 2 years before the study entry,
* stable function of the transplanted kidney during the previous 3 months (changes in s-creatinine ≤ 20%).

Exclusion criteria:

* age less than 18 years,
* symptomatic heart failure,
* malignancy,
* pregnancy or lactation,
* acute conditions and diseases that can affect the GFR,
* newly-introduced drugs that may affect the function of the graft,
* treatment with trimethoprim-sulfamethoxazole or cimetidine,
* the presence of a pacemaker or any other electronic device in the body.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study included 100 kidney transplant recipients (KTRs) with at least 3 months of stable kidney graft function established with estimated GFR (eGFR) according to CKD Epidemiology Collaboration equations, serum creatinine concentration (CKD-EPI Cr), serum cystatin C concentration (CKD-EPI CysC) and measured GFR with 51Cr-EDTA clearance.
  Evaluation of kidney graft function was subject to previous, already completed, and published study (Borštnar Š, et al. Clin Nephrol. 2019;92(6):287-292. doi:10.5414/CN109882). Serum samples from patients participating in this study (taken at the moment of 51Cr-EDTA clearance measurement) were further analyzed in the contemporary study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Association of miRNA and kidney graft function | sample collection within one month of enrollement
  correlation of selected miRNAs expression with parameters of kidney graft function

SECONDARY OUTCOMES:
Association of miRNAs expression and kidney graft rejection or disease recurrence | 2 years
  Correlation of selected miRNAs expression and kidney graft rejection or disease recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No